CLINICAL TRIAL: NCT06409260
Title: Objective Neuromuscular Monitoring in Children (6 Months - 2 Years) With Electromyography and Acceleromyography: A Randomized Study
Brief Title: Neuromuscular Monitoring in Children (6 Months - 2 Years) With Electromyography and Acceleromyography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matias Vested (Other)
Responsible Party: Sponsor-Investigator, Matias Vested, Principal Investigator, Medical Doctor, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMG vs AMG
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: Randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N. tibialis (Other): Objective neuromuscular monitoring done on n. tibialis bilaterally
  Interventions: Other: Acceleromyography (AMG); Other: Electromyography (EMG)
- N. ulnaris (Other): Objective neuromuscular monitoring done on n. ulnaris bilaterally
  Interventions: Other: Acceleromyography (AMG); Other: Electromyography (EMG)

INTERVENTIONS:
Other: Acceleromyography (AMG) — Philips IntelliVue NMT Module
Other: Electromyography (EMG) — Senzime TetraGraph

SUMMARY:
The aim of this study is to compare AMG and EMG (Philips IntelliVue NMT module and Senzime TetraGraph) in the objective monitoring of neuromuscular blocking in children between the age of 6 months and 2 years.The monitoring will be done bilaterally either on n.ulnaris or n. tibialis. The hypothesis of the study is that AMG will indicate faster recovery time (time to return to TOF 90%) from neuromuscular block than EMG.

DETAILED DESCRIPTION:
Objective neuromuscular monitoring is strongly recommended when administering neuromuscular blocking agents (NMBA). However, objective neuromuscular monitoring may be challenging, especially in smaller children due to the limited size of their extremities which often are not easily accessible due to issues such as sterile draping and surgical equipment. Consequently, paediatric anaesthesia care providers often experience problems with neuromuscular monitoring.

NMBAs improve intubating conditions and prevent airway injury in children and infants (<12 months of age). However, both patient age and type of anaesthesia influence onset and duration of action. Infants have shorter onset time of NMBAs compared to older children, and a higher proportion of infants had excellent intubating conditions compared to older children at two minutes after a dose of 0.15 mg/kg cisatracurium. Inhalation anaesthetics prolong recovery from cisatracurium compared to total intravenous anaesthesia and a longer duration of action is seen in infants compared to older children. However, as compared to adults, less profound neuromuscular blockade may be sufficient in children to establish satisfactory intubating conditions.

In children < 3 years old, a study reported residual neuromuscular blockade (TOF (Train Of Four) ratio < 0.9) among 8% of the included patients after administration of a single bolus of 0.1 mg/kg cisatracurium, but the actual proportion may have been as high as 20%. To prevent residual neuromuscular block, objective neuromuscular monitoring is recommended. In adults residual neuromuscular block may result in respiratory events (hypoxaemia and airway obstruction), unpleasant symptoms of muscle weakness, prolonged post-anaesthesia care unit stay, and an increased risk of postoperative pulmonary complications.

It is possible to monitor onset time and duration of action of NMBAs with electromyography (EMG) or acceleromyography (AMG) by train-of-four (TOF) stimulation of a peripheral nerve. Typically, the ulnar nerve is stimulated. In smaller children the tibial nerve can be used as an alternative. However, a recent study in adults reports that there may be important differences when comparing EMG and AMG TOF monitoring at the ulnar nerve with EMG detecting recovery of neuromuscular function later than AMG. Only one study in infants has reported that monitoring of neuromuscular function with AMG applied on the first toe may be a suitable alternative when the thumb is inaccessible. One recent study has reported the feasibility of monitoring the depth of neuromuscular block in infants using electromyography. No study has to our knowledge compared AMG to EMG in infants and small children.

The investigators hypothesize that AMG will indicate faster recovery (time to return to TOF 90%) from neuromuscular block than EMG A secondary aim of this study is to investigate agreement between the two monitors using a Bland Altman analysis comparing onset time and recovery from deep to moderate rocuronium-induced neuromuscular block with EMG and AMG.

ELIGIBILITY:
Inclusion Criteria:

* Patients 6 months - 2 years of age
* Scheduled for elective surgery under general anaesthesia with intubation and use of rocuronium
* American Society of Anesthesiologists (ASA) physical status classification I to III

Exclusion Criteria:

* Known allergy to rocuronium
* Neuromuscular disease that may interfere with neuromuscular data
* Indication for rapid sequence induction
* Prone position

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Time from injection of rocuronium until appearance of the first TOF ratio ≥ 90 | 12 Hours
  Duration of action, defined as time from end of injection of rocuronium 0.6 mg/kg (2xED95) until appearance of the first TOF (Train Of Four) ratio ≥ 90% monitored at the tibial or ulnar nerve.

SECONDARY OUTCOMES:
Bland Altman analysis | Within 12 Hours
  Agreement between the EMG and AMG monitors using a Bland Altman analysis comparing onset time and recovery from deep to moderate NMB with EMG and AMG
TOFC=0 | Within 1 Hour
  Time to TOF-Count=0
TOFR ≥ 0.90 | Within 4 Hours
  Time to TOFR ≥ 0.90

OTHER OUTCOMES:
TOFC=2 | Within 2 Hours
  Time to TOF-Count =2
Control TOF | Within 1 Hour
  Control TOF ratio (baseline) before administration of rocuronium
First PTC | Within 1 Hour
  Time to reappearance of the first response of PTC (PTC=1)
First TOF=1 | Within 1 Hour
  Time to reappearance of the first response to TOF (TOFC=1)
Final TOFR | Within 12 hours
  Final TOF ratio (defined as the TOF ratio upon conclusion of anesthesia)
Difference between control and final TOFR | Within 12 Hours
  Difference between control and final TOF ratio
AMG-TOF ratio when EMG-TOFR ≥ 0.90 | Within 12 Hours
  AMG-TOF ratio when EMG-TOFR ≥ 0.90
EMG-TOF ratio when AMG-TOFR ≥ 0.90 | Within 12 Hours
  EMG-TOF ratio when AMG-TOFR ≥ 0.90
Number of artefacts | Within 12 Hours
  Numbers of artefacts defined as appearance of ≥ one twitch with amplitude of ≥ 5% height in a period of ≥ 30 seconds with TOF 0
Residual neuromuscular blockade | Within 1 hour postoperatively
  Signs and symptoms of residual neuromuscular blockade
  * dysphagia/ swallowing impairment assessed by observing difficulties swallowing (yes/no) or
  * upper airway obstruction
  * desaturation defined as more than 2 minutes with spO2 < 93%
  * reintubation

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested, Study Chair — Rigshospitalet University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No